CLINICAL TRIAL: NCT00644553
Title: A Phase IIIB/IV Comparative Study of the Safety and Efficacy of Clarithromycin Extended-Release Tablets vs. Amoxicillin-Clavulanate for the Treatment of Subjects With Acute Bacterial Sinusitis
Brief Title: Comparative Study of the Safety and Efficacy of Clarithromycin Extended-Release Tablets Versus Amoxicillin-Clavulanate for the Treatment of Acute Bacterial Sinusitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Angela M Nilius, PhD, Abbott
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M02-524
Record Dates: First submitted 2008-03-22; First posted 2008-03-27 (Estimated); Last update posted 2008-03-27 (Estimated); Status verified 2008-03

CONDITIONS: Acute Bacterial Sinusitis (ABS)
MeSH Terms: interventions — Clarithromycin; Amoxicillin; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Clarithromycin
- B (Active Comparator)
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Clarithromycin — Clarithromycin Extended-Release 500 mg tablet (2 tablets QD)
  Other Names: ABT-268; Biaxin
  Arms: A
Drug: Amoxicillin — Amoxicillin-clavulanate 875/125 mg tablet (1 tablet BID)
  Other Names: amoxicillin-clavulanate
  Arms: B

SUMMARY:
To compare the safety/tolerability and efficacy of a 14-day course of clarithromycin extended-release tablets (2 x 500 mg QD) with that of a 14-day course of amoxicillin-clavulanate tablets (875/125 mg BID) for the treatment of ambulatory subjects with Acute Bacterial Sinusitis (ABS).

ELIGIBILITY:
Inclusion Criteria:

* The female must be non-lactating and at no risk for pregnancy.
* Subject must have a diagnosis of ABS. The diagnosis must be based on the following:

  * A sinus radiograph (Water's view) or CT scan with evidence of maxillary opacification or
  * Air/fluid levels purulent discharge from the nose
  * At least two of the following additional signs and symptoms lasting longer than seven days prior to and no longer than 28 days before Evaluation 1.
  * A pre-treatment sample from a sinus puncture or
  * Middle meatus endoscopy must be obtained for bacterial aerobic culture
  * Susceptibility testing (applicable only for selected investigative sites).
* Subject must be a suitable candidate for oral antibiotic therapy and able to swallow tablets intact.

Exclusion Criteria:

* A medical history of hypersensitivity or allergic reactions to clarithromycin, erythromycin, amoxicillin/clavulanate, any penicillin or any of the macrolide antibiotics.
* History of amoxicillin-clavulanate associated cholestatic jaundicehepatic dysfunction.
* Females who are pregnant or lactating.
* Subject has either of the following:

  * Chronic sinusitis (signs and symptoms lasting longer than 28 days immediately prior to Evaluation 1)
  * Significant anatomical abnormalities of the sinuses any other infection or
  * Condition which necessitates use of a concomitant systemic antibiotic.
* Evidence of uncontrolled clinically significant cardiovascular, pulmonary, metabolic, gastrointestinal, neurological, psychiatric or endocrine disease, malignancy, or other abnormality (other than the disease being studied).
* Any underlying condition/disease, that would be likely to interfere with the completion of the course of study drug therapy or follow-up.
* Known significant renal or hepatic impairment (or disease).
* Subject who has taken: a systemic antibiotic within 2 weeks before study drug administration or a long-acting injectable antibiotic (e.g., penicillin G benzathine) within 4 weeks before study drug administration.
* Immunocompromised subjects (e.g., neutropenic subjects).
* Subjects with known HIV infection.
* Treatment with any other investigational drug within 4 weeks prior to study drug administration.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2003-05; Primary Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Clinical Response | 33 days

SECONDARY OUTCOMES:
Radiographic Response | 33 days

CONTACTS AND LOCATIONS:
Locations (44):
- United States (12):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Clovis, California
  - La Jolla, California
  - San Luis Obispo, California
  - Coeur d'Alene, Idaho
  - Charlotte, North Carolina
  - Columbus, Ohio
  - Eugene, Oregon
  - Johnson City, Tennessee
  - San Antonio, Texas
  - Spokane, Washington
- Canada (4):
  - Kitchener, Ontario
  - Toronto, Ontario
  - Sherbrooke, Quebec
  - Saskatoon, Saskatchewan
- Greece (4):
  - Athens
  - Pátrai
  - Piraeus
  - Thessaloniki
- Hungary (4):
  - Budapest
  - Salgótarján
  - Szombathely
  - Veszprém
- Italy (5):
  - Catania
  - Genova
  - Padua
  - Palermo
  - Pavia
- Lithuania (2):
  - Kaunas
  - Vilnius
- Poland (7):
  - Bialystok
  - Bielsko-Biala
  - Bydgoszcz
  - Gliwice
  - Jelenia Góra
  - Lublin
  - Wroclaw
- Bucharest, Romania
- Spain (5):
  - Badajoz
  - Barcelona
  - Madrid
  - Palma de Mallorca
  - Valladolid